CLINICAL TRIAL: NCT00607009
Title: Email-Based Diet and Activity Promotion in Worksites
Brief Title: Project ALIVE (A Lifestyle Intervention Via Email)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CN-04BSter-02-H; 5R01DP000095-03 (NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): ALIVE - received emails about chosen behavioral intervention path - physical activity, fruits/vegetables or fats/sugars
  Interventions: Behavioral: ALIVE
- Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: ALIVE — ALIVE email-based behavioral program based on the participants selected intervention - physical activity, fats/sugars or fruits/vegetabls
  Arms: Intervention

SUMMARY:
The objective of this study is to test the effectiveness of an email-based diet and physical activity intervention on increasing physical activity and fruit and vegetable consumption and decreasing intake of saturated and trans fats and added sugars.

ELIGIBILITY:
Inclusion Criteria:

* regional Northern California KP employees

Exclusion Criteria:

* none

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2006-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
change in physical activity | 4 months

SECONDARY OUTCOMES:
change in fruits and vegetables | 4 months
health-related quality of life | 4 months
presentism | 4 months
stage of change | 4 months
self efficacy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sternfeld, PhD, Principal Investigator — Kaiser Permanente

REFERENCES:
- [Derived] Sternfeld B, Block C, Quesenberry CP Jr, Block TJ, Husson G, Norris JC, Nelson M, Block G. Improving diet and physical activity with ALIVE: a worksite randomized trial. Am J Prev Med. 2009 Jun;36(6):475-83. doi: 10.1016/j.amepre.2009.01.036. PMID 19460655
- [Derived] Block G, Sternfeld B, Block CH, Block TJ, Norris J, Hopkins D, Quesenberry CP Jr, Husson G, Clancy HA. Development of Alive! (A Lifestyle Intervention Via Email), and its effect on health-related quality of life, presenteeism, and other behavioral outcomes: randomized controlled trial. J Med Internet Res. 2008 Nov 19;10(4):e43. doi: 10.2196/jmir.1112. PMID 19019818
- See also: Prevent diabetes: NutritionQuest's new intervention program, Alive-PD. See Dr. Block's presentation on results of randomized trial — https://www.youtube.com/watch?v=F0j5yTXJRqM&feature=youtu.be&list=PLWIrCndjhuYtC8yHcOQJIRiGrnGvRWHxY&noredirect=1